CLINICAL TRIAL: NCT00812799
Title: A Randomised Double Blind Placebo-controlled, Long-term Phase III Study to Assess the Efficacy and Safety of Oralgen Grass Pollen in Patients With Grass Pollen Related Allergic Rhinoconjunctivitis
Brief Title: A Randomised, Double-blind, Placebo Controlled Study With Oralgen Grass Pollen Rhinoconjunctivitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Artu Biologicals (Industry)
Responsible Party: Dr. F.F. Roossien, Artu Biologicals Europe B.V.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB0801
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: randomised; double-blind; placebo-controlled; efficacy and safety; Oralgen® Grass Pollen; allergic rhinoconjunctivitis; allergy; rhinoconjunctivitis; immunotherapy; grass pollen extract
MeSH Terms: conditions — Hypersensitivity | interventions — grass pollen extract, alum-adsorbed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grass pollen extract (Active Comparator): Subjects will receive 19.000 BU grass pollen extract daily sublingually
  Interventions: Drug: Oralgen
- Placebo control (Placebo Comparator): Subjects will receive matching placebo control daily sublingually
  Interventions: Other: placebo control

INTERVENTIONS:
Drug: Oralgen — 19.000 BU daily
  Other Names: Grass pollen extract
  Arms: Grass pollen extract
Other: placebo control — placebo control
  Arms: Placebo control

SUMMARY:
This study will be performed to determine the long-term efficacy of 19.000 BU Oralgen grass pollen administered daily in patients with grass pollen related allergic rhinoconjunctivitis.

DETAILED DESCRIPTION:
Patients between 18 and 60 years will be randomized to receive either Oralgen grass pollen or placebo administered sublingually once a day. Treatment will start at least 16 weeks prior to the anticipated start of the pollen season 2009 and will last until the end of the pollen season 2011. Study medication will be titrated during the first period of treatment until maintenance dose has been reached.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* grass pollen related rhinoconjunctivitis symptoms for at least the last 2 pollen seasons
* positive skin prick test RRTSS greater or equal to 12 during the 2008 season
* signed informed consent

Exclusion Criteria:

* positive skin prick test for other environmental allergens and suffering from serious allergic symptoms
* clinical history of significant symptomatic allergic rhinitis due to tree/weed pollen which potentially overlap the grass pollen season
* clinical history of symptomatic perennial allergic rhinitis caused by an allergen to which the patient is regularly exposed
* lacking of good health
* abnormal spirometry
* lower respiratory tract infection
* asthma requiring treatment other than beta-2 agonists
* oral steroids within 12 weeks before screening
* regular contraindications for use of immunotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Difference between active and placebo-group based on combined RTSS and RMS score | third season

SECONDARY OUTCOMES:
Difference between active and placebo based on RTSS score | third season

CONTACTS AND LOCATIONS:
Overall Officials: Folkert Roossien, Study Director — Artu-Biologicals Europe B.V.
Locations (60):
- Belgium (6):
  - AZ St Jan, Campus Sint-Jan, Bruges
  - Clinique Saint Luc, Brussels
  - U.Z. St Raphael, Leuven
  - University Hospital Leuven, Leuven
  - CHR de la Citadelle, Liège
  - Clinique UCL de Mont-Godinne, Yvoir
- France (9):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Gael Taburet, Brest
  - Francois Durand Perdriel, Nantes
  - Francois Wessel, Nantes
  - Michel Anton, Nantes
  - Françoise Sanquer, Quimper
  - Bruno Lebeaupin, Rezé
  - CHRU de Strasbourg, Strasbourg
  - Mathieu Larrousse, Toulon
- Germany (10):
  - Allergie-Centrum-Charité, Berlin
  - Berufsgen. kliniken Bergmannsheil, Bochum
  - Universitätsklinik Bonn, Bonn
  - Uniklinikum Carl Gustav Carus, Dresden
  - Uniklinikum Frankfurt, Frankfurt am Main
  - MedicoKIT, Goch
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum der Universität München, München
  - Universitätsklinikum Münster, Münster
- Netherlands (6):
  - Rijnland Ziekenhuis, Location Alphen - Poli KNO, Alphen aan den Rijn
  - Wilhelmina ziekenhuis, Assen
  - Ampha De Bilt, De Bilt
  - Catharina Ziekenhuis, Eindhoven
  - AMPHA Nijmegen, Nijmegen
  - Sint Elisabeth Ziekenhuis, Tilburg
- Poland (11):
  - Prywatna Praktyka Lekarska, Gabinet Pediatryczno Alergologiczny, Bialystok
  - SP-ZOZ Osrodek Zdrowia w Bienkowce, Bieńkówka
  - SPZOZ Wojewodzki Szpital Kliniczny im.Dr.J.Biziela, Bydgoszcz
  - Slaskie Centrum Osteoporozy, Katowice
  - SP ZOZ Uniwersytecki Szpital Kliniczny Nr 1, Lodz
  - NZOZ Centrum Alergologii Prof. Buczylko, Lodz
  - SPZOZ Wojewodzki Szpital Specjalistyczny im. Stefana Kardynała Wyszyńskiego, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - NZOZ Lekarze Specjalisci, Wroclaw
  - Szpital Kliniczny Nr 1 im. Prof. Stanislawa Szyszko Slaskiego Uniwersytetu Medycznego w Katowicach, Zabrze
  - Samodzielny Publiczny Szpital Kliniczny nr 3, Zabrze
- United Kingdom (18):
  - The Alverton Practice, Penzance, Cornwall
  - Saltash Health Centre, Saltash, Cornwall
  - Cape Cornwall Surgery, St Just, Cornwall
  - Fowey River Practice, Fowey, Cornwal
  - Sea Road Surgery, Bexhill-on-Sea, Past Sussex
  - Atherstone Surgery, Atherstone, Warwickshire
  - The Porch Surgery, Corsham, Wiltshire
  - Layton Medical Centre, Blackpool, Lancashire
  - Brighton General Hospital, Brighton
  - Hathaway Medical Centre, Chippenham
  - House Surgery, Crownhill, Plymouth
  - Guy's Hospital, Guy's and St Thomas' NHS Foundation Trust, London
  - St. Mary's Hospital, London
  - Royal National Throat, Nose & Ear Hospital, London
  - QMC Notthingham, Nottingham University Hospitals NHS Trust, Nottingham
  - Brannel Surgery, Saint Stephen, Saint Austell
  - Northern General Hospital, Sheffield
  - Avenue Surgery, Warminster